CLINICAL TRIAL: NCT07369258
Title: Music to Prevent Delirium: A Prospective, Randomized, Controlled, Three-Arm Parallel-Group Clinical Trial in an Argentine Intensive Care Unit
Brief Title: Clinical Application of Listening to Music to Prevent Delirium in the Intensive Care Unit
Acronym: CALM-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HOSPITAL BRITANICO DE BUENOS AIRES (Other)
Responsible Party: Principal Investigator, Sebastián Consalvo, Principal Investigator, HOSPITAL BRITANICO DE BUENOS AIRES
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15667
Record Dates: First submitted 2026-01-15; First posted 2026-01-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Critical Illness; Delirium
Keywords: Music; Intensive Care Units; Non-pharmacological Interventions; Psychomotor Agitation; Aged; Music Listening; ICU Delirium; RASS; CAM-ICU
MeSH Terms: conditions — Critical Illness; Delirium; Psychomotor Agitation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Three-arm parallel-group randomized controlled trial with a 1:1:1 allocation ratio
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention (music via headphones), blinding of participants and care providers is not feasible. However, the Outcome Assessor responsible for the daily CAM-ICU and RASS evaluation is blinded to group assignment. To ensure blinding, music devices are not present in the patient's room during the assessment and intervention delivery is recorded in separate study forms (CRFs) rather than the routine medical chart to prevent unblinding via chart review.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Patients receive the institutional Standard of Care (ABCDEF Bundle) for delirium prevention. Participants and families are asked to avoid the use of music devices during the fixed 7-day study window; however, music use is not actively prohibited if requested by the patient or occurs using personal devices. Any such exposure is recorded as protocol deviation ("contamination"), including estimated duration (minutes), source, and type of exposure.
  Interventions: Other: Standard of Care
- Relaxing Music (Experimental): In addition to Standard of Care, patients receive 30-minute music sessions twice daily (morning/afternoon) for up to 7 days after randomization. The playlist consists of standardized, slow-tempo (60-80 bpm) instrumental tracks without lyrics.
  Interventions: Other: Relaxing Music; Other: Standard of Care
- Personalized Music (Experimental): In addition to Standard of Care, patients receive 30-minute music sessions twice daily (morning/afternoon) for up to 7 days after randomization. The playlist consists of songs selected by the patient or proxy based on personal preferences to evoke positive emotions.
  Interventions: Other: Personalized Music; Other: Standard of Care

INTERVENTIONS:
Other: Personalized Music — Delivery of music via circumaural headphones (approximately 60-70 dB; comfortable, non-excessive volume). Playlists are curated based on patient or proxy interviews reflecting prior music preferences. Sessions last at least 30 minutes, twice daily, for up to 7 days after randomization.
  Arms: Personalized Music
Other: Relaxing Music — Delivery via circumaural headphones (approximately 60-70 dB; comfortable, non-excessive volume). Standardized, non-lyrical instrumental tracks (60-80 bpm) designed to induce relaxation. Sessions last at least 30 minutes, twice daily, for up to 7 days after randomization.
  Arms: Relaxing Music
Other: Standard of Care — Institutional standard of care based on the ABCDEF Bundle for ICU patients: (A) Assess, prevent, and manage pain; (B) Both Spontaneous Awakening Trials (SAT) and Spontaneous Breathing Trials (SBT); (C) Choice of analgesia and sedation; (D) Delirium: Assess, prevent, and manage (including daily monitoring via CAM-ICU); (E) Early mobility and exercise; (F) Family engagement and empowerment. Additionally, participants in this group are permitted to access usual environmental media (e.g., television, spoken-word radio, news) as part of routine care.

SUMMARY:
The goal of this clinical trial is to learn if listening to music can prevent delirium in older adults admitted to the Intensive Care Unit (ICU). The main questions it aims to answer are:

* Does listening to music increase the number of days participants are alive and free of delirium and coma during a 7-day period?
* Is personalized music more effective than generic relaxing music?

Researchers will compare Personalized Music and Relaxing Music to Standard Care (no study-provided music) to see if the music intervention improves delirium outcomes compared to usual care.

Participants will:

* Listen to music through headphones twice daily (morning and afternoon) for at least 30 minutes during a 7-day period (intervention groups).
* Receive standard ICU care and undergo daily assessments for delirium and level of consciousness.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Delirium is a prevalent form of acute brain dysfunction in the Intensive Care Unit (ICU), affecting a significant proportion of older critically ill adults, including those receiving invasive mechanical ventilation. It is independently associated with increased mortality, long-term cognitive impairment, and higher healthcare costs. Current pharmacological strategies for delirium prevention have limited efficacy; consequently, clinical guidelines recommend multicomponent non-pharmacological interventions. This study aims to evaluate the clinical effectiveness of a structured music listening intervention as a preventive strategy in older ICU patients.

STUDY DESIGN AND SETTING This study is a single-center, prospective, randomized, controlled trial with three parallel groups conducted in the mixed medical-surgical Intensive Care Unit (27 beds) at the Hospital Británico de Buenos Aires, Argentina.

RECRUITMENT AND RANDOMIZATION Patients admitted to the ICU are screened daily. To ensure inclusion of high-acuity patients (including those receiving invasive mechanical ventilation), screening continues until the patient becomes evaluable. The recruitment window opens during the first 24 hours after the patient first achieves an adequate level of consciousness (RASS -2 to +2) and is confirmed CAM-ICU negative. Randomization must occur within 24 hours of the patient first becoming evaluable and no later than 120 hours (5 days) from ICU admission. Patients who are CAM-ICU positive are not eligible for randomization. Patients who do not become evaluable within 120 hours of ICU admission are not eligible. Allocation is managed via a secure, web-based automated randomization module (REDCap) hosted on the Hospital Británico server. To ensure allocation concealment, the sequence is generated by an independent statistician using permuted blocks of random sizes and loaded into the system. The assignment is revealed to the investigator only after the participant's baseline data has been entered into the system.

INTERVENTION PROTOCOL The protocol consists of music sessions scheduled twice daily in two predefined time windows (Morning: 08:00-12:00; Afternoon: 14:00-20:00) to allow controlled delivery without interfering with ICU care. Each session lasts at least 30 minutes for up to 7 days after randomization, and the first session is started ideally within 2 hours (maximum 4 hours) after randomization unless clinically contraindicated or delayed by procedures. All protocolized sessions are delivered exclusively using study-provided MP3 players and circumaural headphones to ensure technical standardization. Outside the protocolized sessions, participants may listen to additional music using either study equipment or personal devices, with source and minutes recorded separately. Research staff perform a visual check 15 minutes into each session to support protocol fidelity. Sessions may end before 30 minutes if delirium develops (e.g., agitation) or at the participant's request. Study staff ensure that the volume is comfortable and not excessively loud (approximately equivalent to normal conversation, 60-70 dB). Headphones and MP3 players undergo cleaning/disinfection per institutional Infection Control standards between patients. Minutes of total music exposure are recorded daily. In the Relaxing Music arm, any listening that is not consistent with the assigned relaxing-music intervention is recorded as a protocol deviation ("contamination"), with minutes documented. Personalized Music (MP): Playlists are curated based on the participant's prior music preferences (songs provided for loading onto the study MP3 player) and aim to evoke positive emotions. Relaxing Music (MR): Standardized playlists feature slow-tempo (60-80 bpm) instrumental tracks without lyrics. Intervention delivery and daily outcome assessment cease at the earliest of day 7, documented ICU transfer order, death, or withdrawal of consent.

CONTROL GROUP AND STANDARD OF CARE The Control arm receives the institutional standard of care for delirium prevention (ABCDEF Bundle). Importantly, this standard of care is provided to all study participants regardless of group assignment. To preserve the integrity of the comparison, Control participants and families are asked to avoid using music devices during the fixed 7-day study window; however, music is not actively prohibited if the patient requests it or uses personal equipment. Any such exposure is recorded as a protocol deviation ("contamination"), including duration (minutes) and type of exposure. Television or spoken-word radio (e.g., news, podcasts) is allowed as part of usual care.

BLINDING AND ASSESSMENT Delirium assessment is performed daily by a blinded investigator unaware of group assignment. The assessment integrates direct observation using CAM-ICU and a structured chart review of nursing notes from the previous 24 hours using a predefined delirium chart-review algorithm (Chart Review method). The routine blinded assessment is performed daily at 12:00 (±2 hours). Any positive assessment (in-person CAM-ICU or Chart Review) classifies that calendar day as a delirium day (non-free day). To reduce misclassification due to sedatives/analgesics, CAM-ICU assessment is deferred until at least 2 hours after a sedative/analgesic bolus or discontinuation of a continuous infusion.

PRIMARY ENDPOINT (OPERATIONAL DEFINITION) The primary endpoint is Days Alive and Free of Delirium and Coma (DCFDs; range 0-7) in a fixed 7-day window starting on the calendar day of randomization (day 1). Coma days are defined as RASS -3, -4 or -5 and are considered non-free days (CAM-ICU is not performed on coma days). If a participant receives a medical discharge order (transfer order) from the ICU before day 7, remaining days are considered free days (regardless of physical discharge delays); if death occurs before day 7, remaining days are considered non-free days.

KEY SECONDARY ENDPOINT DEFINITIONS While full secondary outcomes are listed in the specific data fields, the following operational definition is specified to distinguish it from the primary endpoint logic: ICU Length of Stay (ICU LOS): Defined as the duration from ICU admission until physical discharge from the unit (actual transfer out of the ICU). Unlike the primary endpoint (DCFDs), which uses the documented medical transfer order to define ICU discharge for endpoint adjudication (regardless of physical discharge delays), ICU LOS captures the total duration of ICU bed occupancy, including administrative delays, to reflect resource utilization.

SAMPLE SIZE ASSESSMENT A total of 330 participants is planned (1:1:1 allocation; 110 per arm). Sample size was defined to ensure adequate power for the primary confirmatory objective under a hierarchical gatekeeping strategy, assuming a minimally clinically relevant difference of 1 day in the primary endpoint (DCFDs) with a common standard deviation of 2.5 days and a two-sided alpha of 0.05, using an asymptotic normal approximation as a conservative reference. The pre-specified primary confirmatory comparison is Combined Music (MP+MR; n=220) versus Control (n=110), providing >90% power under these assumptions. The theoretical reference size for a 1:1 comparison is approximately n≈99 per group for 80% power (relevant for MP vs MR to detect a 1-day difference). The final planned size (110 per arm) includes a 10% increase over the theoretical reference to account for missing data within the 7-day evaluation window and preserve ITT power. Because DCFDs is discrete and bounded (0-7) and the confirmatory test is non-parametric (Mann-Whitney U), the normal-approximation sizing is considered conservative; where appropriate, a simulation-based check under plausible DCFDs distributions may be performed as an internal robustness assessment.

STATISTICAL ANALYSIS PLAN AND GATEKEEPING The primary analysis follows the Intention-to-Treat (ITT) principle. The primary endpoint (DCFDs, 0-7) will be compared using a two-sided Mann-Whitney U test (Wilcoxon rank-sum). Results will be reported as medians [IQR]. Effect size will be reported using the Hodges-Lehmann shift estimate with 95% confidence intervals, and a probability-of-superiority measure (e.g., Cliff's delta or an equivalent estimator) will be provided to facilitate clinical interpretation. To control the global type I error rate and address the clinical questions in a pre-specified priority order, a hierarchical gatekeeping strategy is employed (two-sided alpha=0.05): Step 1 (Confirmatory): Combined Music (MP + MR) versus Control for DCFDs. Step 2 (Key Secondary, under gatekeeping): Performed only if Step 1 is statistically significant (p<0.05); MP versus MR for DCFDs, using the same two-sided Mann-Whitney U test (alpha=0.05). Sensitivity and consistency analyses are pre-specified. Because Mann-Whitney is unadjusted, a sensitivity analysis using robust regression (or quantile regression) will adjust for pre-specified baseline covariates (age, APACHE II, and baseline invasive mechanical ventilation) to confirm robustness to chance baseline imbalances; however, the unadjusted Mann-Whitney test remains the primary basis for confirmatory conclusions. Independently of the gatekeeping outcome, individual comparisons (MP vs Control and MR vs Control) will be reported descriptively with point estimates and 95% confidence intervals as consistency analyses. Secondary outcomes will be interpreted as exploratory, except for two key supportive endpoints (incidence of delirium and days with delirium), for which Holm-Bonferroni adjustment will be applied within that predefined family (family-wise alpha=0.05); supportive endpoints do not determine confirmatory conclusions.

MISSING DATA Proactive procedures (daily monitoring, eCRF alerts, and redundancy via chart review) are implemented a priori with the goal of keeping missingness below 5%. Missing data handling for DCFDs is pre-specified and follows the operational definition of the endpoint. Days with RASS ≤ -3 are classified as coma (non-free days) without requiring CAM-ICU. For evaluable days (RASS ≥ -2) with missing CAM-ICU, the primary ITT analysis uses Multiple Imputation by Chained Equations (MICE) with a longitudinal multilevel approach (including a subject-level random effect), generating m ≥ 20 imputed datasets. Predictors include baseline variables (e.g., age, APACHE II, baseline invasive mechanical ventilation), available daily measures (e.g., RASS, sedation dose), and prior-day status. DCFDs is derived within each imputed dataset and combined using Rubin's rules. Sensitivity analyses include complete-case analysis if overall missingness is <5% and a conservative worst-case scenario imputing all missing evaluable days as non-free (delirium positive).

SUBGROUP AND EXPLORATORY ANALYSES A pre-specified subgroup analysis evaluates heterogeneity of treatment effect in participants receiving invasive mechanical ventilation (IMV) at baseline using a Group × Baseline IMV interaction term adjusted by APACHE II. For time-to-event outcomes in ventilated participants (time to successful extubation), death is treated as a competing risk; the primary analysis uses a Fine-Gray competing risks model (subdistribution hazard ratio, sHR), with a cause-specific Cox model as sensitivity analysis. A pre-specified landmark sensitivity analysis at 4 hours post-randomization will be performed, restricting to participants who remain mechanically ventilated at that time; additional landmark thresholds between 2 and 6 hours will be evaluated as sensitivity analyses. Ventilator-free days at 28 days (VFD-28) will be compared using Mann-Whitney U due to its composite distribution. An exploratory dose-response analysis will assess the association between total music minutes (continuous) and DCFDs within the intervention arms using robust regression (or quantile regression), adjusting for baseline severity (APACHE II) and a sedation-depth indicator (e.g., average RASS), recognizing potential confounding by illness severity and reverse causality; results will be interpreted as exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older.
* Negative Confusion Assessment Method for the ICU (CAM-ICU) at the time of randomization.
* Expected ICU length of stay of at least 48 hours based on clinical judgement at admission (e.g., need for mechanical ventilation, vasopressors, invasive monitoring).

Exclusion Criteria:

* Positive CAM-ICU prior to randomization.
* Acute primary Central Nervous System pathology (e.g., ischemic or hemorrhagic stroke, traumatic brain injury, meningoencephalitis, intracranial hypertension) presenting with altered sensorium (Glasgow Coma Scale at admission < 14) or focal deficit preventing cognitive assessment (e.g., severe aphasia).
* Severe chronic cognitive impairment or advanced dementia, defined by a known history of severe functional dependence prior to admission (requiring permanent assistance for basic activities of daily living such as feeding or grooming)
* Unresolved auditory or visual impairment.
* Suspected or confirmed intoxication with drugs or alcohol at admission.
* Uncontrolled psychiatric disease (at least one acute episode requiring intervention in the last 6 months).
* Richmond Agitation-Sedation Scale (RASS) score < -2 or > +2 at the time of randomization.
* Medical condition precluding the safe use of headphones (e.g., burns, skull fracture, skin lesions).
* Inability to establish effective communication due to a language disorder or unresolved language barrier.
* Inability of the patient or legal representative to provide informed consent.
* Patients with imminent death, end-of-life care, or limitation of therapeutic effort.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Days Alive and Free of Delirium and Coma | From randomization up to Day 7
  Number of days alive and free of delirium and coma (range 0-7) in a fixed 7-day window (Day 1 = calendar day of randomization). Coma is defined as a Richmond Agitation-Sedation Scale (RASS) score of -3 to -5 (scale range: +4 [combative] to -5 [unarousable]). Delirium is defined as the presence of delirium assessed by the Confusion Assessment Method for the ICU (CAM-ICU) or by a positive chart review (screening nursing notes for delirium-related keywords); CAM-ICU is not assessed during coma. Assessments are performed daily. A day is "free" only if the patient is alive, has RASS ≥ -2, and is delirium-negative on both CAM-ICU and chart review. ICU discharge order (transfer order) before Day 7: remaining days counted free. Death before Day 7: remaining days counted non-free. Higher values indicate better outcomes.

SECONDARY OUTCOMES:
Days with Delirium | From randomization up to Day 7
  Number of delirium-positive days in a fixed 7-day window (Day 1 = calendar day of randomization), assessed daily on days with RASS ≥ -2. A delirium-positive day is defined as any day with a positive CAM-ICU assessment and/or a positive structured chart review of nursing notes (Chart Review method; screening for delirium-related keywords). If multiple assessments occur within a day and any is positive, that calendar day is counted as a delirium day.
Days with Coma | From randomization up to Day 7
  Number of coma days in the fixed 7-day window (Day 1 = calendar day of randomization). Coma = RASS -3, -4 or -5. CAM-ICU not assessed during coma.
Incidence of Delirium | From randomization up to Day 7
  Proportion of participants with at least one delirium-positive day during the fixed 7-day window (Day 1 = calendar day of randomization), assessed daily on days with RASS ≥ -2. A delirium-positive day is defined as any day with a positive CAM-ICU assessment and/or a positive structured chart review of nursing notes (Chart Review method; screening for delirium-related keywords). Reported by group as the proportion with ≥1 delirium day.
Mortality During Intervention | From randomization up to Day 7
  Occurrence of death from any cause within the 7-day intervention window after randomization (Yes/No).
Intensive Care Unit Length of Stay | From ICU admission to physical ICU discharge, assessed up to 90 days
  Total duration of stay in the Intensive Care Unit calculated from admission to physical discharge
Cumulative Antipsychotic Load | From randomization up to Day 7
  Total cumulative antipsychotic dose during Days 1-7, converted to chlorpromazine equivalents and expressed as mg/kg using actual body weight at ICU admission (pre-specified conversion table).
Cumulative Benzodiazepine Load | From randomization up to Day 7
  Total cumulative benzodiazepine dose during Days 1-7, converted to lorazepam equivalents and expressed as mg/kg using actual body weight at ICU admission (pre-specified conversion table).
Cumulative Dexmedetomidine Load | From randomization up to Day 7
  Total cumulative dexmedetomidine during Days 1-7, expressed as μg/kg using actual body weight at ICU admission (sum of infusion rate × duration).
Cumulative Opioid Load | From randomization up to Day 7
  Total cumulative opioid dose during Days 1-7, converted to oral morphine equivalents and expressed as mg/kg using actual body weight at ICU admission (pre-specified conversion table).
Cumulative Propofol Load | From randomization up to Day 7
  Total cumulative propofol dose administered during Days 1-7, expressed as mg/kg using actual body weight at ICU admission (includes bolus doses and continuous infusions).
Change in Anxiety Level | From randomization up to Day 7 (assessed twice daily)
  Numeric Rating Scale (NRS) 0-10 (0=no anxiety, 10=worst possible anxiety) in communicable participants (RASS -2 to +2). Assessed immediately before and within 10 minutes after each music session. Outcome is per-session change (post minus pre).
Days with Physical Restraints | From randomization up to Day 7
  Number of days (0-7) in which the patient required physical restraints due to psychomotor agitation; a day counts if restraints were used at any time during that day.
Time to Successful Extubation | From randomization until successful extubation, assessed up to ICU discharge or Day 90, whichever occurs first
  Time from randomization to successful extubation, defined as 48 hours without reintubation and without need for noninvasive ventilatory support. Analyzed in participants receiving invasive mechanical ventilation at randomization; censored at ICU discharge (per protocol definition) or at Day 90.
Ventilator-Free Days at Day 28 | From randomization up to Day 28
  Number of days alive and free of invasive mechanical ventilation during the 28 days after randomization (range 0-28); participants who die before Day 28 are assigned 0.

OTHER OUTCOMES:
Total Music Exposure | From randomization up to Day 7
  Total minutes of music listening accumulated per participant during Days 1-7 (sum of protocolized sessions and any additional non-protocolized listening), recorded daily in the study CRFs.
Percentage of Completed Sessions | From randomization up to Day 7
  Percentage of scheduled sessions that were fully completed (defined as >= 30 minutes of uninterrupted listening)
Incidence of Ear Injury | From randomization up to Day 7
  Presence of pressure ulcers or skin injury on the ear auricle caused by headphone use (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastián Consalvo, MD, Principal Investigator — Hospital Británico de Buenos Aires
Locations (1):
- Hospital Británico de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided
A formal data sharing plan is not yet in place. Currently, data access is restricted to the research team as per the approved protocol. Future sharing may be considered upon reasonable request subject to ethics committee approval